CLINICAL TRIAL: NCT06466096
Title: Correlation Analysis of Postoperative Delirium and Postoperative Neurocognitive Disorder in Elderly Patients With Gastrointestinal Neoplasms
Brief Title: Correlation Analysis of POD and pNCD in Elderly Patients With Gastrointestinal Neoplasms
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 27961988
Record Dates: First submitted 2024-06-03; First posted 2024-06-20 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Delirium; Postoperative Neurocognitive Disorder; Gastrointestinal Surgery
Keywords: postoperative delirium; postoperative neurocognitive disorder; serum indicators; gastrointestinal neoplasms surgery
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- postoperative delirium(POD) and postoperative neurocognitive disorder(pNCD): Delirium (CAM scale ) was assessed 7 days after surgery and divided into POD and non-POD groups; one of the above scenarios indicated postoperative delirium;The patients in the POD group were evaluated for cognitive function at 1 month and 12 months after surgery to determine whether pNCD occurred. The patients in the POD group were further divided into pNCD subgroup and non-PNCD subgroup, and the changes of serum indicators before and after surgery in the pNCD and non-pNCD subgroups were compared.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — this is an observation study, no intervention

SUMMARY:
This is a prospective cohort study to explore the differences of serum indicators between elderly gastrointestinal neoplasms patients with postoperative delirium (POD) who either develop or do not develop long-term postoperative neurocognitive disorders (pNCD).

DETAILED DESCRIPTION:
The purpose of this study is to explore the differences of serum indicators between elderly gastrointestinal neoplasms patients with postoperative delirium (POD) who either develop or do not develop long-term postoperative neurocognitive disorders (pNCD).

Elderly gastrointestinal neoplasms patients aged 65 and above, undergoing surgical operations at Xuanwu Hospital, Capital Medical University, were selected. The serum indicators of all patients were measured before surgery, and neurocognitive function of all patients was assessed using the Montreal Cognitive Assessment (MoCA) within 1 week before surgery. General patient data such as sex, age, comorbidities, BMI, ASA classification, and MoCA scores were collected. Under routine anesthetic management of the Department of Anesthesiology and Surgical Operations at Xuanwu Hospital, endotracheal intubation general anesthesia was performed. Intraoperative monitoring included heart rate, blood pressure, pulse oximetry, and body temperature, with surgery and anesthesia times, and fluid balance recorded. The serum indicators of all patients were measured after surgery. Within 7 days post-surgery, delirium assessment was conducted using the Confusion Assessment Method (CAM), classifying patients into POD and non-POD groups. For the patients in the POD group, neurocognitive function was assessed at a period of time after surgery to determine the presence of pNCD, further dividing the POD group into pNCD and non-pNCD subgroups. The correlation between POD and pNCD was explored by comparing the changes of serum indicators before and after surgery in the pNCD and non-pNCD subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥65 years of age who have undergone surgical anesthesia of gastrointestinal neoplasms; Sign informed consent.

Exclusion Criteria:

* Inability to complete cognitive function assessment; Illiteracy, hearing impairment or visual impairment; He has a history of epilepsy, depression, schizophrenia, Alzheimer's disease and other psychiatric and neurological diseases.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients 65~100 years of age who have undergone surgical anesthesia of gastrointestinal neoplasms
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
the changes of blood biomarkers before and after surgery between elderly gastrointestinal neoplasms patients with postoperative delirium (POD) who either develop or do not develop postoperative neurocognitive disorders (pNCD) one month after surgery | 2024.5.9-2026.6.1
  Perioperative changes in blood-based biomarkers can reflect the pathophysiological processes of diseases. Current studies indicate that the perioperative levels of blood-based biomarkers may be associated with postoperative neurocognitive disorders in elderly patients. These blood-based biomarkers may provide novel avenues for the early diagnosis, prevention, and improvement of outcomes in elderly patients with postoperative neurocognitive disorders.
  The procedures are as follows:
  Neurocognitive function assessments were conducted on the enrolled patients within one week before surgery, one month after surgery, and twelve months after surgery, respectively. Whether the patients developed postoperative delirium was evaluated within seven days after surgery. Venous blood was drawn before surgery and within three days after surgery to detect the levels of brain-derived neurotrophic factor (BDNF), high-sensitivity C-reactive protein (hs-CRP), and homocysteine (Hcy).

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No